CLINICAL TRIAL: NCT06452836
Title: Colors, Can They Reduce the Dental Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SelcukU004
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Anxiety State; Tooth Extraction Status Nos
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Translucent Glasses Group (Placebo Comparator)
  Interventions: Other: control
- Green Colored Glasses Group (Experimental)
  Interventions: Other: Green color exposure
- Red Colored Glasses Group (Experimental)
  Interventions: Other: Red color exposure
- Blue Colored Glasses Group (Experimental)
  Interventions: Other: Blue color exposure

INTERVENTIONS:
Other: Green color exposure — Patients will wear green colored glasses before and during the surgery.
  Arms: Green Colored Glasses Group
Other: Red color exposure — Patients will wear red colored glasses before and during the surgery.
  Arms: Red Colored Glasses Group
Other: Blue color exposure — Patients will wear blue colored glasses before and during the surgery.
  Arms: Blue Colored Glasses Group
Other: control — Patients will wear translucent glasses before and during the surgery.
  Arms: Translucent Glasses Group

SUMMARY:
The investigator's aim in this study was to evaluate the preoperative anxiety and pain felt during the operation due to exposure to green, red, and blue light. For this purpose, the participants will wear colored glasses before the operation. The investigator will evaluate the patient's anxiety change and the pain she/he feels during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and ASA 2 patient population
* not having had a third molar surgery before
* volunteer to participate in the study

Exclusion Criteria:

* dental phobia
* patients who will be treated under general anesthesia
* refusing the measurements
* not filling out the VAS
* encountering complications during surgery
* operations lasting more than 45 minutes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Anxiety Score | 1 minute after the participant sits the dental unit and 10 minutes after
  Patients fill out the Dental Anxiety Scale(Visual Analogue Scale) when they sit in the dental unit. Ten minutes after the glasses are worn, patients fill out the anxiety scale again. Changes in the scores are the primary outcome of the study. The scale range is 0-10. A lower score means better results.

SECONDARY OUTCOMES:
Change in the oxygen saturation | 1 minute after the participant sits the dental unit and 10 minutes after
  Saturation measurement is done from the fingertip using a pulse oximeter one minute after the patient sits in the dental unit and after ten minutes. Changes in the scores are the secondary outcome of the study. The average value is above %90.
Change in the pulsation | 1 minute after the participant sits the dental unit and 10 minutes after
  Pulsation was measured from the fingertip by a pulse oximeter one minute after the patient sat in the dental unit and after ten minutes. Changes in the scores are the secondary outcome of the study. The average value is between 65 and 75.
Intraoperative Pain Score | 1 minutes after the surgery
  Measuring the pain felt by the patient after the operation with the help of the visual analog scale. The range of Scala is 0-10. A lower score means better results.
Change in the salivary cortisol level | 1 minute after the participant sits the dental unit and 10 minutes after
  Measuring the salivary cortisol level one minute after the patient sits in the dental unit and after ten minutes. Changes in the levels are the secondary outcome of the study.
Change in the salivary alfa-amilase level | 1 minute after the participant sits the dental unit and 10 minutes after
  Measuring the salivary alfa-amylase level one minute after the patient sits in the dental unit and after ten minutes. Changes in the levels are the secondary outcome of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Gürses, Study Chair — Selcuk University, Faculty of Dentistry; İsmail Okumuş, Principal Investigator — Selcuk University, Faculty of Medicine
Locations (1):
- Selcuk University, Faculty of Dentistry, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided